CLINICAL TRIAL: NCT04038905
Title: The Use of Digital Genetic Counselor (DGC) for BRCA1/2 Mutation Carrier Testing
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Igentify Ltd (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 007250
Record Dates: First submitted 2019-07-28; First posted 2019-07-31 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2019-07

CONDITIONS: BRCA Mutations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The DGC provides an end-to-end solution to the Oncogenetics screening process from participant registration to receipt of the genetic test results and their interpretation. These steps are provided using personalized animated videos.

DETAILED DESCRIPTION:
Step 1. Registration: During the initial phone call with potential participants, qualified staff that are part of the study will explain the process and extend an invitation to participated in the study. The DGC process will begin when the Sheba MC Genetics Institute will send potential participants a link. Participant will undergo the standard two-factor authentication method based on phone number and last four digits of the ID number. At the end of this process a new user will be created in the system. Note: There are no physical risks associated with participation in this study.

Step 2. Interactive medical questionnaire: The interactive medical questionnaire is defined as the process of gathering personal information relevant to the specific clinical genetic scenario (e.g. personal information, personal and family medical information). The questionnaire is dynamic and is interactively adapted based on live information supplied by the participant. The questionnaire was approved by the Sheba MC PI.

Please note that the essence of the DGC system is to enable to conduct genetically relevant medical informatics processes in the context of digital sessions with secured and adaptive systems.

One of the major aims of the questionnaire is to enable the use of the scientific risk calculator "BRCAPRO" (a breast and ovarian cancer risk assessment algorithm accepted by Israel MOH). This allows the DGC to provide the participant with her risks for being a BRCA mutation carrier and the risk of developing breast/ovarian cancer prior to the oncogenetic test.

At the end of that phase of the DGC use, the participant will be informed that: "You are presented with a questionnaire regarding genetic test for having a mutation in BRCA1/2, by answering the questions you hereby accept the participation this medical questionnaire. Before the submission of DNA sample to the test you will be asked to sign an Informed Consent for the participation in the study, that this questionnaire is part of it." Note: The genetic test is part of a routine test performed at the Sheba MC Genetic Institute and is not part of this study. Participants will be asked to sign the routine Informed Consent for the genetic test.

Step 4. Sample submission and signing a hard copy Informed Consent for the BRCA1/2 test: At the Sheba MC Genetic Institute, before the submission of buccal/saliva/blood samples to the test, participants will be asked to sign a hard copy Informed Consent.

Step 5. Introductory personalized animated video: A personalized and dynamic animated video is machine-generated following a well-characterized medically supervised algorithm to tailor the video to each participant. The algorithm that generates the personalized introductory video is approved by the Sheba medical staff. Participants will receive a short-animated video summarizing the medical process they are going through, the potential risks and other details that they need to know and understand before approving and continuing with the procedure. The content of these videos is dynamic and in full alignment with the Sheba MC requirements.

The dynamic video is generated by a third party that receives ONLY the following information:

1. Participant first name
2. Participant age
3. Is the participant having one of the following cancers: breast, ovarian, pancreas, stomach, uterus or other. As a general approach we need to address women with cancer differently than cancer free women. In addition, the potential risks of breast and ovarian cancers is different. The pancreas, stomach, uterus indications are important as identification of a mutation in the BRCA1/2 genes may lead to change in the therapeutic options for these women.
4. Is the risk for harboring a mutation in BRCA1/2 as determined by BRCAPRO 10% or above?
5. Is the risk for breast cancer according BRCAPRO greater than 20%?

Following the dynamic video, the system will examine participants' understanding by a short interactive quiz that summarizes the relevant topics presented in the video. Following the quiz, the participant will be asked to sign an electronic Informed Consent for carrying out the routine mutation carrier test in the BRCA1/2 genes. When the participants come to the Genetics Institute to provide the buccal/saliva/blood samples, she will re-sign a hard copy of the Informed Consent in front of the clinician. It is important for the usability study to test the responsiveness of the participant to sign the electronic Informed Consent following the personalized introductory video.

The investigators believe that this video will provide a clear and, in most cases, more thorough explanation than the common face-to-face explanation.

On Board Dashboard for the Medical Staff: A dedicated dashboard enables medical staff to monitor the advancement of a participant throughout the process. It will include all the information gathered from the participant through the on-line registration and questionnaire and a genetic counselor is able to revise the data. The genetic counselor can send the participant a signed summary letter (PDF) via the secure DGC system and invite him/her to perform the genetic test. Following completion of data entering of the medical questionnaire, the system will automatically run the BRCAPRO risk calculator to predict the participant predicted lifetime risk of having breast cancer and of being a BRCA1/2 gene mutation carrier. In case the risk for harboring a mutation in the BRCA1/2 genes is 10% or higher, the cost of the genetic test is reimbursed by the HMO (in the "health basket"). In those cases, the participant will receive a signed letter summarizing her family history and specifying the calculated risk for carrying a BRCA mutation to enable HMO reimbursement of the test cost (TOFES 17). For women where the estimated risk for harboring mutation is less than 10% the cost of the test is out of pocket for the participant.

Once the participant concludes the session of Participant Enrollment (Pre-Test), all her data are presented in the medical staff dashboard. A genetic counselor will be able to edit the data mainly derived from the self-reported questionnaire and the BRCAPRO predictions. Next, the genetic counselor will send the participant a signed summary letter (PDF) via the DGC system. This letter will present the information entered into the system by the participant and invite her to perform the genetic test. Using the standard two-factor authentication method based on phone number and the last four digits of the participants' ID number, the participants will be able to view the report. In cases of risk harboring a mutation in the BRCA genes >10% that qualify with reimbursed by the HMO, the letter to the participant will also include the information how to ask for HMO reimbursement.

Counseling logic - the logics of the DGC system (the "brain"):

DGC Algorithm: The results of the genetic test chosen by the health care providers are uploaded to the Sheba MC system via an interface for this specific genetic test. Next, the system utilizes its medically-supervised genetic algorithm to decide on the outcome of the genetic counseling. The algorithm takes advantage of all relevant information in the system including the predictions of the risk calculator BRCAPRO. The outcomes of the system are either a digital genetic counseling report generator (see next section) or an invitation to a face-to-face genetic counseling session to receive the results. All women who are found to harbor a germline mutation in the BRCA1/2 genes will be invited to a face-to-face genetic counseling session.

Risk Calculators: Provide evidence-based estimation of the risk of the participant to develop Breast Cancer and Ovarian cancer as well as to be carrier of a mutation in the BRCA1/2 genes. As mentioned above, risk calculations using a variety of algorithms can be performed before and after the genetic test. Pretest calculations are done in order to see if risks justify by law HMO coverage of the genetic test. Post-test run of the calculators aims to provide the residual risk taking into account the results of the genetic test. The BRCAPRO algorithm is based on posterior calculations of residual carrier risk, genetic test results, ethnicity, and pre-existing knowledge of carrier state frequencies in the given population.

Interface for genetic results: In the current study, the DGC will work only with the results of the test done at the Sheba MC Oncogenetic laboratory for the 14 BRCA1/2 mutations prevalent in Israeli population.

Counseling Summary Session:

This module is responsible to generate two types of outputs. Low risk participants (namely individuals that based on their personal and family history in conjunction with the test results are deemed at a low risk of having an inherited predisposition to cancer) are approved to receive an automated digital report (personalized video), while high risk participants are urged to schedule a face-to-face genetic counseling session. In high risk cases, the genetic counselor will have the digital information provided by the participants and the genetic test results, to make the counseling process more effective. The threshold of High/Low risk assignment is determined by the head of the head of Sheba MC Genetic Institute.

Digital Genetic Counseling Report Generator: This component generates an animated, personalized dynamic video and a written report (in PDF format) summarizing the genetic counseling provided to the participant online. The report is machine-generated and approved by medical personnel before its disclosure to the participant. Using the standard two-factor authentication method based on phone number and the last four digits of the participants' ID number, the participants will be able to view the personalized video and download the reports.

Support for face-to-face Genetic Counseling: The system dashboards will present the genetic counselor with a full report containing all gathered information to-date, augmented with digital tools, such as animated videos aimed to facilitate an effective session.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to undergo BRCA1/2 genotyping
* Participants willing to use the DGC as part of their genetic screen
* Participants willing to fill up follow up questionnaires about their experience and understanding of the genetic counseling, and share their clinical and DGC usage data with the study personnel
* Fluent in Hebrew
* Age 18 or above

Exclusion Criteria:

* Individuals that underwent bone marrow transplantation.
* Participants refusing to participate in the study.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Israeli female
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in number of face-to-face pre-test and post-test genetic counseling sessions | One year
  The investigators expect that the pre-test session of all participants will be handled using the enrollment module of the system making the face-to-face session unneeded. In addition, the investigators expect that about 10% of BRCA negative, low risk women that received digital counseling will still request a face-to-face counseling session. Overall, the investigators estimate that the 55% of the women will not require a post-test face-to-face session.

CONTACTS AND LOCATIONS:
Overall Officials: Elon Pras, Prof., Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No